CLINICAL TRIAL: NCT02865655
Title: Cesarean Section Scar Evaluation by Saline Contrast Sonohysterography During Hysteroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiFMIH-CSD
Record Dates: First submitted 2016-08-10; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Cesarean Section Scar
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- CSD-TVU: Cesarean Section Scar Evaluation by TVU
- CSD-MRI: Cesarean Section Scar Evaluation by MRI
- CSD-MRI with saline: Cesarean Section Scar Evaluation by MRI with saline
- CSD-Hysteroscopic: Cesarean Section Scar Evaluation by Saline Contrast Sonohysterography During Hysteroscopy
  Interventions: Procedure: Hysteroscopic

INTERVENTIONS:
Procedure: Hysteroscopic
  Groups: CSD-Hysteroscopic

SUMMARY:
To apply an existing diagnostic imaging test (saline infusion sonohysterography by Hysteroscopic) to characterize the "filling defect" of a previous cervical cesarean delivery scar in the nonpregnant uterus

ELIGIBILITY:
Inclusion Criteria:

cesarean section diverticula patients in our hospital from 2016 to Dec 2018.The diagnosis was confirmed on the basis of medical history (at least one C-section), clinical symptoms (post¬menstrual spotting, no significant change of cycle before and after C-section),transvaginal ultrasonography (TVU), and mag¬netic resonance imaging (MRI) findings

Exclusion Criteria:

1) irregular menstrual cycle before cesar¬ean section; 2) previous placement of an intrauterine contracep¬tive device; and 3) presence of another organic uterine pathology responsible for abnormal uterine bleeding examined by hysteroscopy, such as endome-trial hyperplasia, endometrial polyps, malignancy, or submucosal myomas

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: cesarean section diverticula patients in our hospital from 2016 to Dec 2018.The diagnosis was confirmed on the basis of medical history (at least one C-section), clinical symptoms (post¬menstrual spotting, no significant change of cycle before and after C-section),transvaginal ultrasonography (TVU), and mag¬netic resonance imaging (MRI) findings
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Cesarean Section Scar Evaluation by TVU and MRI | 2015.12-2016.7

CONTACTS AND LOCATIONS:
Overall Officials: Xipeng Wang, Study Chair — Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University
Locations (1):
- Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University, Shanghai, Shanghai Municipality, China